CLINICAL TRIAL: NCT05368402
Title: Randomized, Placebo-controlled, Double-blinded, 2-parallel Arm, Clinical Trial Evaluating Ladarixin 400 mg Bid as Adjunctive Therapy to Improve Glycemic Control in Overweight Insulin-resistant Patients With Type 1 Diabetes.
Brief Title: Clinical Trial on Ladarixin Adjunctive Therapy to Improve Glycemic Control in Type 1 Diabetes.
Acronym: CONSERVA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low recruitment rate
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LDX0122; 2022-000743-68 (EudraCT Number)
Record Dates: First submitted 2022-05-05; First posted 2022-05-10 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Type 1 Diabetes
Keywords: glycemic control; insulin-resistant type 1 diabetes.
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — 2'-((4'-trifluoromethanesulfonyloxy)phenyl)-N-methanesulfonylpropionamide

STUDY DESIGN:
Intervention Model Description: Patients across all genders, 21-65 years, inclusive, with established insulin-requiring T1D and IR, will be assigned (1:1) to receive either oral ladarixin 400 mg b.i.d. for 7 cycles (26 weeks) of 14 days on/14 days off (treatment group) or matched placebo (control group) for a total of 28 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Appearance, including packaging and labelling, of the IMP (capsules, packaging) will not allow to recognize actual treatment (either ladarixin or placebo).
  During the trial, blinding will be broken by the Investigator for emergency purposes only, where knowledge of the blinded treatment could influence further patient care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ladarixin (Experimental): Ladarixin was administered orally at the dose of 400 mg b.i.d. for 7 cycles of 14 days with an interval of 14 days off, for a total duration of 26 weeks.
  Interventions: Drug: Ladarixin
- Placebo (Placebo Comparator): Matching placebo was administered with the same treatment schedule of the IMP.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ladarixin — The two daily oral doses of ladarixin (400 mg each dose) were administered at about a 12-hour interval (morning and evening; ideally between 6:30/11:30 and 18:30/23:30). At each administration, 2 capsules were swallowed with a glass of water, at least 2 hours apart from breakfast or dinner
  Other Names: LDX
  Arms: Ladarixin
Other: Placebo — Placebo was administered with the same ladarixin schedule.
  Arms: Placebo

SUMMARY:
Primary objective

- To determine whether oral ladarixin versus placebo adjunctive therapy improves glycemic control in overweight, insulin resistant (IR) adult subjects with type 1 diabetes (T1D).

Secondary objectives

* To ascertain the effect of ladarixin on glycemic variability as per CGM derived parameters.
* To determine the safety of oral ladarixin versus placebo adjunctive therapy in overweight, IR adult subjects with T1D.

DETAILED DESCRIPTION:
This study is a randomized, placebo-controlled, double-blinded, 2- parallel arm, phase II trial.

The planned number of patients to be enrolled was 86, across all genders, 21-65 years, inclusive, with established insulin-requiring T1D and IR, to be assigned (1:1) to receive either oral ladarixin 400 mg b.i.d. for 7 cycles (26 weeks) of 14 days on/14 days off (treatment group) or matched placebo (control group).

The planned duration of treatment was 7 cycles of 14 days with an interval of 14 days off (no IMP), for 26 weeks and a for total of 5 study visits.

Actually, only 24 patients were screened, 3 enrolled and 2 were randomized. The study was terminated early due to low recruitment rates; 2 patients completed the study, and therefore only their safety data are relevant to this study report.

No efficacy evaluation was conducted due to small numbers and early study termination. As a result, no conclusions can be made about the effectiveness of the treatment.

Only safety evaluations were conducted: no missing data on safety variables for the 2 randomized participants. At study termination, no TEAEs, ADRs, TESAEs, serious or severe ADRs had occurred, and therefore the safety profile of ladarixin had not changed.

ELIGIBILITY:
Inclusion Criteria:

1. clinical diagnosis of autoimmune T1D as documented by positive T1D-related autoantibodies [the presence of at least one or more of Insulin autoantibodies (IAA), Anti-GAD (GAD65), Anti-IA2 (IA2), Zinc Transporter 8 (ZnT8)];
2. age 21-65 years, inclusive, at the time of consent;
3. T1D duration > 1 year;
4. detectable fasting C-peptide as per the result of screening laboratory measurement;
5. current insulin standard of care (ISOC), either established use of an insulin pump (closed loop system excluded) or a stable dose level and dose frequency for the last two months prior to screening, with no plans to switch the modality of insulin administration during the trial;
6. routine use of a self-owned (if applicable) Continuous Glucose Monitoring (CGM) system that can record glucose concentrations continuously for at least 7 days;
7. HbA1c value >7.5% as per the result of screening laboratory measurement;
8. evidence of IR based on a total daily insulin dose >0.8 U/kg/day;
9. subject is overweight or obese as per body mass index (BMI) of between 24-33 kg/m2, inclusive;
10. ability to comply with all protocol procedures for the duration of the study, including scheduled follow-up visits and examinations, and willing to be contacted by clinical trial staff;
11. provision of signed informed consent prior of any study-related procedure not part of standard medical care.

Exclusion Criteria:

1. use of a "closed loop system" for integrated glucose reading/insulin infusion;
2. known or suspected hypersensitivity to the active pharmaceutical ingredient, non-steroidal anti-inflammatory drugs or any excipient of the investigational medicinal products (e.g. lactose and croscarmellose) as well as patients with congenital lactase deficiency, galactosaemia or glucose-galactose intolerance will have to be excluded;
3. use of non-insulin medications for adjunctive blood glucose control (e.g: antidiabetic agents such as metformin, sulfonylureas, glinides, thiazolidinediones, exenatide, liraglutide, DPP-IV inhibitors, SGLT-2 inhibitors or amylin) within one month of randomization as well as required in the participant's standard of care;
4. use of medications for weight reduction such as: Belviq (lorcaserin), Qsymia (Phentermine + topiramate), Orlistat (xenical) within one month of randomization as well as required in the participant's standard of care;
5. use of a medication such as stimulants, antidepressants and/or psychotropic agents that could affect weight gain or glycemic control of T1D;
6. treatment with drugs metabolized by CYP2C9 with a narrow therapeutic index [i.e., phenytoin, warfarin, and high dose of amitriptyline (>50 mg/day)];
7. use of angiotensin-converting enzyme inhibitors, interferons, quinidine antimalarial drugs, lithium, niacin;
8. evidence of QTcF >470 msec and a history of significant cardiovascular disease/abnormality;
9. any condition, including unstable diet and disordered eating behaviour, that in the judgment of the investigator will adversely affect patient's safety or the completion of the protocol or otherwise confound study outcome;
10. pregnancy (subjects of child-bearing potential) based on serum test (quantitative beta hCG) at screening; unwillingness to use effective contraceptive measures up to 2 months following trial discharge (all participants);
11. clinical diagnosis of celiac disease that is in poor control as defined by most recent tissue transglutaminase (tTG) that is in the abnormal range;
12. history of ≥1 Diabetic Ketoacidosis (DKA) events in the past 6 months;
13. hypoalbuminemia (serum albumin <3 g/dL);
14. hepatic dysfunction defined by increased ALT/AST > 3 x upper limit of normal (ULN) and increased total bilirubin > 3 mg/dL [>51.3 μmol/L];
15. moderate to severe renal impairment calculated by estimated Glomerular Filtration Rate (eGFR) <60 mL/min/1.73 m2 as determined using Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine equation;
16. past (within 1 month prior to screening) or current administration of any immunosuppressive medications (including oral or systemically injected steroids) and use of any investigational agents, including any agents that impact the immune response;
17. a condition already known which interferes with the ability to accurately determine glycated HbA1c;
18. significant systemic infection during the 4 weeks before the 1st dose of study drug (e.g., infection requiring hospitalization, major surgery, or i.v. antibiotics to resolve; other infections, e.g., bronchitis, sinusitis, localized cellulitis, candidiasis, or urinary tract infections, must be assessed on a case-by-case basis by the investigator regarding whether they are serious enough to warrant exclusion).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Pozzilli, MD, Principal Investigator — Campus Bio-Medico di Roma (UCBM) Policlinico Universitario, Rome, Italy, 00128
Locations (2):
- Italy (2):
  - Ospedale F. Spaziani Frosinone, Frosinone
  - Università Campus Bio-Medico di Roma (UCBM) Policlinico Universitario, Rome

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 24 participants who were screened, 21 failed to meet eligibility criteria, and 3 were enrolled, of which 2 were randomized: 1 in the IMP arm and 1 in the placebo arm. The third enrolled participant was not randomized after being enrolled due to study interruption by the sponsor.
Period: Overall Study
Arm/Group | Ladarixin | Placebo
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ladarixin | Placebo | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Italy | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an HbA1c Reduction From Baseline of ≥0.50% (Absolute Difference) Without Episodes of Severe Hypoglycemia.
Description: Please note that this outcome is meant to express the "count" (number + %) of participants. Please also note that because of the low recruitment rate (out of the 24 participants screened, only 2 participants were enrolled, 1 in the ladarixin group and 1 in the placebo group), it was not possible to have a consistent sample size for any formal statistical analyses, accordingly no efficacy evaluation was conducted on the two randomized subjects' data.
  The low recruitment rate led the Sponsor decide to close enrollment on 04th August 2023 and thus to early terminate the study.
Time Frame: At Visit 4 (week 27/28)
Population: There were only two participants recruited in the study e.g., 1 in the Ladarixin group and 1 in the placebo group. Due to the low recruitment rate, the Sponsor decided to close enrollment on 04th August 2023 and thus to early terminate the study.
  Accordingly, Population consists of the two randomized participants only.
Measure: Count of Participants; unit: Participants
Arm/Group | Ladarixin | Placebo
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

2. Secondary Outcome: Number of Patients With Treatment Emergent Adverse Events (TEAEs) of Any Kind From the Beginning of Study Treatment to up to the End of Study Participation
Description: Number of Patients With Treatment Emergent Adverse Events (TEAEs) of Any Kind From the Beginning of Study Treatment administration to up to the End of Study Participation was reported.
  AE= any untoward medical occurrence after exposure to a medicine, which is not necessarily caused by that medicine.
  serious AE (SAE)= any adverse event that results in death, is life-threatening, requires hospitalisation or prolongation of existing hospitalisation, results in persistent or significant disability or incapacity, or is a birth defect.
  non serious AE(nsAE)= any adverse drug experience associated with the use of the Product in humans, whether or not considered drug-related, which is not a Serious Adverse Event.
Time Frame: Throughout the study, up to week 26 (day 182)
Population: randomized patients
Measure: Count of Participants; unit: Participants
Arm/Group | Ladarixin | Placebo
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Throughout the study up to week 26 (day 182), for the only 2 patients with safety results.
Arm/Group | Ladarixin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
On 4th August 2023, the Sponsor decided to close enrollment because of a low recruitment rate (as per Clinical Study Protocol). At that time two patients were randomized out of a total of 24 screened, while 86 patients were expected to be enrolled by December 2022. Given the low recruitment rate, no formal statistical analyses could be undertaken for assess IMP efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/02/NCT05368402/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/02/NCT05368402/SAP_001.pdf